CLINICAL TRIAL: NCT02498886
Title: An Exploratory Study to Determine Bioavailability and Transferrin Saturation Following a Single Dose of a Novel Iron Supplement (IHAT) in Gambian Women.
Brief Title: IHAT Absorption Kinetics
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, dora pereira, Senior Investigator Scientist, Medical Research Council
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 1422
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Iron-deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iron deficient anaemic: IDA (Experimental): Iron deficient anaemic women.
  Interventions: two iron supplements will be used:
  IHAT- iron hydroxide adipate tartrate: an analogue of natural food iron. Ferrous sulphate- the gold standard for iron supplementation. For both the iron single-dose will be 60mg elemental iron equivalent.
  Each compound will be labelled with a stable isotope of iron:
  IHAT with 2 mg 58Fe and ferrous sulphate with 10 mg 57Fe.
  1 capsule of each compound will be ingested with a full glass of water in two separate occasions, 14 days apart.
  Interventions: Dietary Supplement: IHAT; Dietary Supplement: Ferrous sulphate
- Iron sufficient: non-IDA (Experimental): Women that are not anaemic or iron deficient.
  Interventions: two iron supplements will be used:
  IHAT- iron hydroxide adipate tartrate: an analogue of natural food iron. Ferrous sulphate- the gold standard for iron supplementation. For both the iron single-dose will be 60mg elemental iron equivalent.
  Each compound will be labelled with a stable isotope of iron:
  IHAT with 2 mg 58Fe and ferrous sulphate with 10 mg 57Fe.
  1 capsule of each compound will be ingested with a full glass of water in two separate occasions, 14 days apart.
  Interventions: Dietary Supplement: IHAT; Dietary Supplement: Ferrous sulphate
- Iron deficient anaemic (IDA): IHAT new manufacture (Experimental): Iron deficient anaemic women.
  Interventions: two iron supplements will be used:
  IHAT new manufacture- iron hydroxide adipate tartrate: an analogue of natural food iron.
  Ferrous sulphate- the gold standard for iron supplementation. For both the iron single-dose will be 60mg elemental iron equivalent.
  Each compound will be labelled with a stable isotope of iron:
  IHAT with 2 mg 58Fe and ferrous sulphate with 10 mg 57Fe.
  1 capsule of each compound will be ingested with a full glass of water in two separate occasions, 14 days apart.
  Interventions: Dietary Supplement: IHAT; Dietary Supplement: Ferrous sulphate

INTERVENTIONS:
Dietary Supplement: IHAT — Iron hydroxide adipate tartrate (IHAT): Single dose capsule containing IHAT equivalent to 60mg iron with 2 mg isotopically enriched with 58Fe.
Dietary Supplement: Ferrous sulphate — Ferrous sulphate: Single dose capsule containing ferrous sulphate heptahydrate equivalent to 60 mg iron with 10 mg isotopically enriched with 57Fe.

SUMMARY:
At MRC Human Nutrition Research, the investigators have developed an engineered analogue of the ferritin-core for safe and effective iron supplementation. Iron hydroxide adipate tartrate (IHAT) is a tartrate-modified, nano-disperse Fe(III) oxo-hydroxide, formed in an adipate buffer, with similar functional properties and small primary particle size (~2 nm) as the iron found in the ferritin core; it better mimics iron absorption from food than the non-physiological bolus doses of ferrous sulphate currently used.

This exploratory study will test the hypothesis that IHAT has equivalent bioavailability to ferrous sulphate but produces a less harmful post-ingestion rise in transferrin saturation. The design is a 3-arm (IDA, non-IDA and IDA-IHAT new manufacture), crossover, randomised, single-dose study.

Primary endpoint:

Relative bioavailability value of IHAT versus ferrous sulphate. This will be determined from the red blood cell incorporation of isotope-labelled iron 14 days following a single oral dose.

Secondary endpoints:

Serum iron at 0, 2, 4, 6 hours following a single dose of each iron compound. Transferrin saturation at 0, 2, 4, 6 hours following a single dose of each iron compound.

Plasma 58Fe and 57Fe at 0, 2, 4, 6 hours. Pathogen growth using ex vivo assays in serum collected from each subject at 0, 2, 4 and 6 hours following a single dose.

DETAILED DESCRIPTION:
The study's main hypothesis is that IHAT will be bioavailable in pre-menopausal anaemic Gambian women and will lead to a lower serum iron and transferrin saturation increase than an equivalent dose of ferrous sulphate. Furthermore, the investigators hypothesize that IHAT will produce a less harmful post-ingestion rise in transferrin saturation, i.e. the serum collected from subjects following a single dose of IHAT will promote less pathogen growth in ex vivo assays than that collected following an equivalent dose of ferrous sulphate. Finally, based on previous animal data [5], the investigators hypothesize that IHAT absorption will be significantly higher in anaemic women compared to non-anaemic women, and that this will not be the case with ferrous sulphate.

This study is a cross-over, single-dose comparison against ferrous sulphate (standard of care) in anaemic and non-anaemic women. The iron single dosage for both compounds will be 60mg elemental iron equivalent and each compound will be labelled with a stable iron isotope. Outcomes will be: red blood cell incorporation of labelled iron, serum iron, transferrin saturation and pathogen growth in ex vivo serum assays.

Primary objective:

To determine iron bioavailability (i.e. red blood cell incorporation) from a single dose of IHAT versus ferrous sulphate in pre-menopausal Gambian women.

Secondary objective:

To determine serum iron absorption following a single dose of IHAT versus ferrous sulphate in pre-menopausal Gambian women.

To evaluate if a single-dose of IHAT produces a less harmful post-ingestion rise in transferrin saturation and serum iron than ferrous sulphate.

Each compound is labelled with a stable isotope of Fe so that its absorption can be determined from the red blood cell incorporation of the stable isotope 14 days after the single dose. This study is effectively a Phase 0 study (pharmacokinetics) with small numbers and because iron absorption varies from individual to individual, depending on their body iron needs and gastrointestinal digestion issues, it is more accurate to use each study subject as her own control. Therefore, each subject will ingest IHAT on one study day and the active treatment comparator on a separate day. The 2 study visits need to be 14 days apart to allow for red blood cell incorporation of the stable iron isotopes used to label the iron materials. This method is the gold standard to determine relative bioavailability values (RBV) of novel iron compounds (i.e. in relation to ferrous sulphate absorption) and allows an accurate determination of RBV of IHAT that otherwise would not be possible if we used a parallel study design with small numbers.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women apparently healthy (as judged by a study nurse at the screening day) with normal CRP (measured at screening).
* Non-pregnant (will be tested with a rapid pregnancy test) and non-lactating women.
* IDA arm: 9≤Hb≤11 g/dL and ferritin≤ 15 ng/ml
* Non-IDA arm: Hb>11 g/dL and ferritin> 15 ng/ml.

Exclusion Criteria:

* Malaria and other infections
* Severe anaemia (Hb<9 g/dL)
* CRP> 5 mg/L
* Chronic disease
* Currently participating in other iron intervention studies.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability value of IHAT versus ferrous sulphate | 14 days
  This will be determined from the red blood cell incorporation of isotope-labelled iron 14 days following a single oral dose.

SECONDARY OUTCOMES:
Serum iron | 6 hours
  Serum iron will be determined at 0, 2, 4, 6 hours following a single dose of each iron compounds (i.e. on days 1 and 14).
Transferrin saturation | 6 hours
  Tsat will be determined at 0, 2, 4, 6 hours following a single dose of each iron compounds (i.e. on days 1 and 14).
Pathogen Growth | 6 hours
  Pathogen growth will be determined using ex vivo assays in serum collected from each subject at 0, 2, 4 and 6 hours following a single dose of each compound (days 1 and 14).
Plasma iron | 6 hours
  Plasma 58Fe and 57Fe will be determined at 0, 2, 4, 6 hours (on days 1 and 14).

CONTACTS AND LOCATIONS:
Overall Officials: Dora I Pereira, PhD, Principal Investigator — Medical Research Council
Locations (1):
- MRC Unit The Gambia, Keneba, West Kiang, The Gambia

REFERENCES:
- [Background] Pereira DI, Bruggraber SF, Faria N, Poots LK, Tagmount MA, Aslam MF, Frazer DM, Vulpe CD, Anderson GJ, Powell JJ. Nanoparticulate iron(III) oxo-hydroxide delivers safe iron that is well absorbed and utilised in humans. Nanomedicine. 2014 Nov;10(8):1877-86. doi: 10.1016/j.nano.2014.06.012. Epub 2014 Jun 28. PMID 24983890
- [Background] Powell JJ, Bruggraber SF, Faria N, Poots LK, Hondow N, Pennycook TJ, Latunde-Dada GO, Simpson RJ, Brown AP, Pereira DI. A nano-disperse ferritin-core mimetic that efficiently corrects anemia without luminal iron redox activity. Nanomedicine. 2014 Oct;10(7):1529-38. doi: 10.1016/j.nano.2013.12.011. Epub 2014 Jan 4. PMID 24394211
- [Background] Aslam MF, Frazer DM, Faria N, Bruggraber SF, Wilkins SJ, Mirciov C, Powell JJ, Anderson GJ, Pereira DI. Ferroportin mediates the intestinal absorption of iron from a nanoparticulate ferritin core mimetic in mice. FASEB J. 2014 Aug;28(8):3671-8. doi: 10.1096/fj.14-251520. Epub 2014 Apr 28. PMID 24776745